CLINICAL TRIAL: NCT06969924
Title: Real-World Data on the Effects of Cardiac Resynchronization Therapy in Adult Patients With Congenital Heart Disease
Acronym: RECORD-CHD
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Anastasia D. Egorova, MD, PhD, MD, PhD, Leiden University Medical Center
Other Study IDs: 2023-035
Record Dates: First submitted 2025-04-29; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Adult Congenital Heart Disease
Keywords: Adult congenital heart disease; Cardiac resynchronization therapy; ACHD; CRT; Heart failure; HF
MeSH Terms: conditions — Heart Defects, Congenital; Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- ACHD patients with CRT: All participants included in the registry have to have a congenital heart defect, be ≥ 18 years old and have to have a CRT pacemaker or defibrillator
  Interventions: Device: Cardiac resynchronization therapy

INTERVENTIONS:
Device: Cardiac resynchronization therapy — Cardiac resynchronization therapy pacemaker or defibrillator with a transvenous or epicardial systemic ventricle lead

SUMMARY:
This study aims to evaluate the real-world effects of cardiac resynchronization therapy (CRT) in adult patients with congenital heart disease (ACHD). Specifically, it seeks to determine whether CRT improves clinical outcomes in this unique patient population and to identify factors associated with a favorable response to therapy.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) is well-established in acquired heart failure, but evidence in ACHD remains limited. Current guidelines, extrapolated from non-congenital populations, may not fully address the anatomical and electrophysiological complexities in ACHD.

This retrospective cohort study aims to investigate the real-world efficacy and safety of CRT in adult patients with congenital heart disease (ACHD). The study includes consecutive ACHD patients who underwent either de novo CRT implantation or upgrade procedures, starting from January 2014.

The primary objectives are to evaluate changes in QRS duration, systemic ventricular function, and New York Heart Association (NYHA) functional class. The study aims to further examine the impact of CRT in specific ACHD subgroups, including patients with systemic right ventricles (vs. systemic left ventricles), those with non-left bundle branch block (non-LBBB) morphology (vs. LBBB), and those with upgrade procedures (vs. de novo implants).

Data collection is based on retrospective review of electronic health records, including patient demographics, clinical characteristics, device-related procedural details, and follow-up data. Outcomes are assessed using standardized echocardiographic and electrocardiographic measurements, alongside clinical evaluations.

The study aims to provide comprehensive real-world insights into the efficacy and safety of CRT in the diverse ACHD population and to identify predictors of favorable response, ultimately supporting more individualized decision-making in this complex patient group.

ELIGIBILITY:
Inclusion Criteria:

* ACHD patients who underwent CRT implantation

Exclusion Criteria:

* Less than 18 years old on the moment of CRT implantation
* Patient objection to the use of retrospective data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult congenital heart disease patients who received cardiac resynchronization therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
QRS duration | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on the duration (in ms) of the QRS interval on surface ECG
Systemic ventricle function class | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on the echocardiographic functional classification of the systemic ventricle (i.e., normal, mildly reduced, moderately reduced, severely reduced)
NYHA functional class | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on the NYHA functional classification (i.e., Class I, II, III, IV)

SECONDARY OUTCOMES:
Clinical - Mortality | From enrollment through study completion, with an average follow-up duration of 1 year.
  Death from any cause during the study period
Clinical - Heart failure hospitalization | From enrollment through study completion, with an average follow-up duration of 1 year.
  At least one overnight stay with cardiac decompensation as the primary reason for hospitalization
Clinical - CV hospitalization other than HF | From enrollment through study completion, with an average follow-up duration of 1 year.
  At least one overnight stay due to any primary cardiovascular reason, excluding heart failure
Clinical - Urgent heart failure visit | From enrollment through study completion, with an average follow-up duration of 1 year.
  An unplanned medical contact requiring decongestion, but no overnight stay in the hospital
Clinical - Urgent CV visit other than HF | From enrollment through study completion, with an average follow-up duration of 1 year.
  An unplanned medical contact due to any primary cardiovascular reason, excluding heart failure and without overnight stay in the hospital
Clinical - Enlisting for LVAD | From enrollment through study completion, with an average follow-up duration of 1 year.
  Enlisting for left ventricular assist device (LVAD) implantation during the study period
Clinical - Enlisting for HTX | One year after implantation
  Enlisting for heart transplantation (HTX) during the study period.
Clinical - Periprocedurel complications | From enrollment through study completion, with an average follow-up duration of 1 year.
  Any complications occurring during or immediately after the procedure, including but not limited to pneumothorax, infection, bleeding, lead dislodgement, and arrhythmic events.
CIED-related - Threshold systemic ventricular lead | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal change of the minimum pacing threshold required for consistent ventricular capture, measured in volts (V) at a specific pulse width (ms)
CIED-related - Impedance systemic ventricular lead | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal change of the systemic ventricular lead impedance, measured in ohms (Ω), reflecting the integrity of the pacing system and lead-tissue interface.
CIED-related - R-wave sensing systemic ventricular lead | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal change of the R-wave amplitude of the systemic ventricular lead, measured in millivolts (mV), indicating the ability of the system to correctly sense the ventricular depolarization
CIED-related - ICD therapy | From enrollment through study completion, with an average follow-up duration of 1 year.
  Incidence of (in)appropriate ICD therapies, including shock or antitachycardia pacing
Medication - GDMT use | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal change in the use of guideline-directed medical therapy (GDMT) for heart failure, including RAAS inhibitors (ACEi/ARB/ARNI), mineralocorticoid receptor antagonists (MRA), beta-blockers (BB), diuretics, and SGLT2 inhibitors (SGLT2i).
Clinical parameter - weight | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on weight (kg)
Clinical parameter - systolic blood pressure | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on systolic blood pressure (mmHg)
Clinical parameter - diastolic blood pressure | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on diastolic blood pressure (mmHg)
Clinical parameter - heart rate | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on heart rate (beats per minute)
Laboratory parameter - sodium | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on serum sodium (mmol/L)
Laboratory parameter - creatinine | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on serum creatinine (μmol/L)
Laboratory parameter - eGFR | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on estimated glomerular filtration rate (eGFR, ml/min/1.73m2)
Laboratory parameter - NT-proBNP | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on serum NT-proBNP (ng/L)
Laboratory parameter - hs-TnT | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on serum high-sensitivity troponin T concentrations (ng/L)
Echocardiographic parameter - subpulmonary ventricle function class | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on the echocardiographic functional classification of the subpulmonary ventricle (i.e., normal, mildly reduced, moderately reduced, severely reduced)
Echocardiographic parameter - SAVV regurgitant grade | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on the regurgitant grade of the systemic atrioventricular valve, classified as grade I, II, III, or IV.
Echocardiographic parameter - PAVV regurgitant grade | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on the regurgitant grade of the pulmonary atrioventricular valve, classified as grade I, II, III, or IV.
Echocardiographic parameter - sPAP | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on systolic pulmonary artery pressure (sPAP), estimated by echocardiography.
Echocardiographic parameter - IVC diameter | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of CRT on inferior vena cava diameter and its collapsibility during respiration, as assessed by echocardiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center (LUMC), Leiden, South Holland, Netherlands